CLINICAL TRIAL: NCT05462561
Title: Robotic Vascularized Composite Bladder Allograft Transplantation: A Phase 0 (First-in-Human), Single Institutional Study for Deceased-Donor Bladder Transplantation
Brief Title: Vascularized Composite Bladder Allograft Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4B-21-5; NCI-2022-00076 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 4B-21-5 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Neurogenic Bladder; Bladder Dysfunction; Immunosuppression
Keywords: neurogenic bladder; vascularized composite allograft
MeSH Terms: conditions — Urinary Bladder, Neurogenic

STUDY DESIGN:
Intervention Model Description: 5 total:
  * 1 patient will be accrued for feasibility, and monitored for a period of 3 months.
  * If successful, defined as the absence of life-threatening complication, including allograft rejection requiring explantation, and adequate bladder storage, accrual of the remaining 4 patients will ensue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (VCBA) (Experimental): Patients undergo robotic VCBA transplantation.
  Interventions: Other: Quality-of-Life Assessment; Procedure: Robotic Vascularized Composite Bladder Allograft Transplantation

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Robotic Vascularized Composite Bladder Allograft Transplantation — Undergo robotic VCBA transplantation.

SUMMARY:
This phase 0 trial tests the feasibility, functionality, and sustainability of vascularized composite bladder allograft transplantation in treating patients with terminal bladder pathology. A vascularized bladder allograft transplantation may provide a more durable and better-tolerated alternative to standard urinary diversion, which employs bowel. A robotic surgical approach will be employed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To perform a feasibility study of vascularized composite bladder allograft (VCBA) transplantation and demonstrate successful transplantation of a vascularized composite deceased-donor bladder allograft.

SECONDARY OBJECTIVES:

I. To describe the adverse events associated with VCBA transplantation.

II. To describe the immunosuppression regimen for patients undergoing VCBA transplantation.

III. To evaluate allografted bladder functionality (storage and emptying) after transplantation.

OUTLINE:

This study will be the first to report on the feasibility of human bladder transplantation. In the appropriately selected candidate, a vascularized bladder allograft transplantation may provide a more durable and better-tolerated alternative to urinary diversion using the bowel. The objective of this study is to perform successful, safe robotic genitourinary bladder allotransplantation and define the optimal surgical techniques in up to 5 genitourinary patients using standard triple-therapy immunosuppression. A multi-institutional, multidisciplinary Genitourinary Vascularized Composite Bladder Allograft Transplantation Team has been established to address this aim.

Brain dead donors who have met the criteria for Determination of Death will be selected by the Genitourinary transplant team in conjunction with the organ procurement organization (OPO) for the University of Southern California, OneLegacy. The mandatory requirements are family consent for donation. These criteria are standard and are not part of the research question at hand.

A robotic vascularized composite bladder allograft transplantation will be performed, after which patients will be monitored closely as both an inpatient and at serial timepoints after surgery in the outpatient setting.

This is the critical period when most of the surgical complications leading to allografts loss can take place. During this period, VCBA recipients will remain at the Keck USC Urology Step-down Unit for 7 days following the surgery, from where they will be moved to the regular floor. Daily examinations and post-operative ultrasound evaluation will be performed by the urology service to monitor for signs of rejection. The patient will have protocol biopsies as detailed below and during any rejection episodes. Once drug levels are stable and therapeutic and the patient is without complications, the process of discharge with close follow-up will be initiated.

Immediately after surgery, discharge will typically occur 1-3 weeks following transplantation. A detailed explanation of postoperative discharge instructions will be provided by the discharge nurse, social worker, and transplant coordinator and will include: medication dosages and associated adverse effect profiles (the patient will be instructed to record the time of all medications taken); schedule of required laboratory draws; timing of physician follow-up visits; wound care; assessment of urine output; diet; monitoring of blood pressure and temperature; hygiene; dental care; opportunistic infection prevention; use of gloves and masks; activity and exercise; maintaining a nonsmoking environment; driving; child immunization; caring for house pets; and other special instructions. The endpoint is the success of the transplant, measured by adequate blood flow and no signs of complications.

Evaluation of bladder integrity, including urine output, will be an essential component of transplant surveillance. In addition, graft biopsies will be routinely performed at one month after surgery and every 3 months through cystoscopy during the first year, plus whenever clinically indicated. Biopsies are taken from the bladder dome during in-office cystoscopy. Hemostasis is achieved through Bugby electrocautery. This is a common urologic procedure performed in outpatient surgery centers and urology clinics nationwide. The clinical care needs of each patient will likely be individually different after genitourinary transplantation and will thus be adjusted specifically per patient. Daily monitoring of the quality and quantity of urine output is considered clinically particularly relevant for monitoring graft rejection. Briefly, allograft recipients need to visit the transplant clinic staff once a week for the 1st post-operative month, then once every other week for 1 month, then once monthly for 6 months, and thereafter once every 3 months for the management of immunosuppression and assessment of rejection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years.
* Positive history of one of the following:

  * Bladder pathology resulting in poor compliance, recurrent infections, and/or resultant upper tract (kidney and ureteral) pathology, demonstrated by hydronephrosis with resultant kidney disease.
  * Localized, non-metastatic, muscle-invasive or lesser urothelial cell carcinoma of the bladder that requires therapeutic radical cystectomy will be considered only if the patient is already on pre-existing immunosuppression or who are expected candidates for immunosuppression in the near future, and then on a case-by-case basis after thorough evaluation and presentation to institutional tumor board committee. A minority of accrued patients are expected to have bladder cancer as the etiology of their cystectomy.
* Patients that are on pre-existing immunosuppression will be included in this study.
* Patient agrees to comply with the protocol and states a dedication to the immunomodulatory treatment regime.
* Patients must demonstrate appropriate manual dexterity or sufficient assistance at home to perform clean intermittent catheterizations as needed. The patient (or assistant) must demonstrate proficiency in performing clean intermittent catheterization during pre-transplant workup.
* No co-existing medical condition which, in the opinion of the study team, could affect the immunomodulatory protocol, surgical procedure, or functional results (see Exclusion Criteria below). If the condition is amenable to treatment, the study team must agree that said condition should not significantly enhance the surgical risks of genitourinary transplantation. Examples of such medical conditions would include a burden of atherosclerotic disease that would preclude vascular anastomosis, and psychiatric disorders that would preclude reliable adherence to medications.
* No active co-existing psychosocial problems (i.e., alcoholism, drug abuse).
* Negative crossmatch with donor.
* DONOR: Any potential brain dead donor considered for solid organ transplant.
* DONOR: Age 18-65 years.
* DONOR: Stable, meaning no requirement of excessive vasopressors for maintaining blood pressure.
* DONOR: ABO compatibility.
* DONOR: Negative cross-match with recipient.

Exclusion Criteria:

* Positive history of one of the following medical co-morbidities:

  * Human immunodeficiency virus [HIV] (active or seropositive), active hepatitis B or C, viral encephalitis, untreated sepsis, active tuberculosis, viral encephalitis, toxoplasmosis, varicella zoster virus.
  * Conditions that may impact the success of the surgical procedure or increase the risk of postoperative complications including inherited coagulopathies like hemophilia, Von-Willebrand's disease, protein C and S deficiency, thrombocythemia, thallassemia, sickle cell disease.
  * Mixed connective tissue diseases and collagen disorders (can result in poor wound healing after surgery), including:

    * Mixed connective tissue disorder
    * Severe deforming rheumatoid arthritis
    * Infectious, post-infectious, or inflammatory (axonal or demyelinating) neuropathy
    * Ehler-Danlos syndrome
  * Lipopolysaccharidosis or amyloidosis (effects nerve regeneration).
  * Impaired liver function as evaluate by liver function panel, including the presence of hyperbilirubinemia, elevated aspartate aminotransferase/ alanine aminotransferase (AST/ALT), and the presence of secondary coagulopathy, measured by prothrombin, international normalized ratio, and partial thromboplastin time.
  * Severe anemia (hemoglobin < 7 g/dL), leukopenia (WBC < 3 x 10 ^ 9 cell/L), or thrombocytopenia (platelets < 20 x10 ^ 9 cells/L).
* Oncology patient specific:

  * History of any non-urothelial malignancy within the past 5 years, with the exception of non-melanomatous skin cancer and very-low to low risk prostate cancer on active surveillance.
  * History of metastasic malignancy within the past 5 years.
  * History of urothelial carcinoma in patients without pre-existing conditions that require immunosuppression and/or without the expected need for immunosuppression in the future.
* Sensitized recipients; panel reactive antibody (PRA) < 80%, with negative crossmatch to donor and no evidence of donor-specific antibody at time of transplant.
* Patients unable to receive adequate follow-up care and/or unable to receive immunosuppression due to geographic, financial or other reasons.
* Patients with a smoking history who cannot demonstrate smoking cessation for a period of 6 months prior to listing and a desire to abstain from post-operative smoking will be excluded.
* Records of poor medical compliance, documented psychological disorder(s), substance abuse or incomplete psychological clearance.
* Particular attention will be paid to the candidate's compliance and their desire to undergo the offered procedure. While there is no "score" on any particular evaluation that would rule out a patient, certain factors can aid in the identification of patients who for example may not have the ability to comply with the medical directives necessary to care for a genitourinary transplant, or psychologically are not prepared for transplant, or who have unrealistic expectations about the transplant. The decision on eligibility is a team decision. All members of the team will discuss each candidate in a multidisciplinary meeting and reasons for concern over eligibility will be discussed at a Selection Committee Meeting (per University of Southern California Transplant Center Policy). In circumstances where the candidate is considered to be less suitable, they could be given an opportunity to address these issues either through individual counseling or further education and then be reconsidered as a potential candidate. Every effort to prevent a request for allograft removal will be made. Towards these ends, a two-part initial psychiatric consultation will be rendered in addition to psychosocial evaluations already accounted for in the social work and transplantation evaluation prior to listing. The first visit focuses on background history and standard contraindications to transplantation, while the second visit is a more thorough discussion of the challenges ahead for the potential recipient and how these challenges relate to their strengths and vulnerabilities. If at this phase, or any subsequent one, significant psychological need emerges, the patient will be referred to another mental health professional for ongoing treatment with frequent communication between that provider and the transplant psychiatrist. The same psychiatrist responsible for listing and taking part in the protocol will not provide this treatment, given the potentially conflicting obligations involved and the disincentive present for the patient to be completely honest. If a greater than 6 month period of time elapses between listing and transplantation, a follow-up visit with psychiatry and social work will be arranged.
* DONOR: Unresolved sepsis.
* DONOR: Known history of urothelial or prostate cancer/malignancy.
* DONOR: Known history of bladder or prostate surgery.
* DONOR: Abnormal bladder capacity.
* DONOR: Active sexually transmitted disease.
* DONOR: Active cytomegalovirus (CMV), Epstein-Barr virus (EBV), or tuberculosis (TB) infections.
* DONOR: Hepatitis B virus (HBV) core antibody, surface antigen, or DANN positive.
* DONOR: Hepatitis C virus (HCV) antibody or viral load+.
* DONOR: Human immunodeficiency virus (HIV)/acquired immunodeficiency syndrome (AIDS).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-10-03 (Estimated); Study Completion 2028-10-03 (Estimated)

PRIMARY OUTCOMES:
Technical success of vascularized composite bladder allograft (VCBA) transplantation | At completion of transplantation procedure
  Defined as appropriate vascularization of the transplanted bladder, measured through intraoperative fluorescence imaging and immediate post-operative computed tomographic angiography.

SECONDARY OUTCOMES:
Adverse events associated with VCBA transplantation | Immediately peri-operative and 30 and at 90 days after transplantation
  Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5 criteria will be used to describe adverse events. A rejection episode managed medically will be defined as a grade 3 adverse event, while rejection requiring allograft explanation will be graded as a CTCAE grade 4 event.
Transplant rejection | Up to 1 year within 7 days post-transplantation
  Rejection will be graded using a modified histological grading system adapted from Banff criteria, similar to that adopted in uterine transplantation.
Bladder function | At 7, 30, 90, 180, and 360 days
  Defined by measurements of bladder capacity. The 30 and 90 day timepoints will include cystoscopic evaluation and the 90 day timepoint urodynamic evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Inderbir Gill, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States